CLINICAL TRIAL: NCT00368771
Title: A Six-Month Study to Compare Outcome Differences and Visceral Response in Subjects Randomized to a Psychological Intervention for Irritable Bowel Syndrome
Brief Title: A Six-month Study to Compare Outcome Differences and Visceral Response ... Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NR007768 (NIH); R01NR007768 (NIH); DK-NR07768
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Abdominal Pain; Abdominal Discomfort; Diarrhea; Constipation; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Diarrhea; Constipation

ARMS (3):
- 1 (Active Comparator): IBS Stress Management
  Interventions: Behavioral: IBS Stress Management
- 2 (Active Comparator): IBS Symptom Management
  Interventions: Behavioral: IBS Symptom Management
- 3 (Active Comparator): IBS Educational Training
  Interventions: Behavioral: IBS Educational Training

INTERVENTIONS:
Behavioral: IBS Stress Management — If randomly assigned to this intervention, the session with the therapist will consist of training about IBS symptoms and their relationship to stress, as well as skills training in relaxation and ways of identifying and challenging mistaken thoughts about life events. The goal of this treatment is to lessen mental and physical stressful reactions to daily events, and therefore lessen IBS symptoms as a reaction to stress. The patient will be encouraged to apply relaxation skills to stressful situations.
  Arms: 1
Behavioral: IBS Symptom Management — If assigned to this group, the therapist will discuss feelings, over-attention to IBS symptoms, and your fear of IBS symptoms. Patients will learn how to identify thoughts that may increase your IBS symptoms and will practice how to change these thoughts to ones that make them feel more comfortable. The sessions will focus on reactions to daily life that in turn result in IBS Symptoms.
  Arms: 2
Behavioral: IBS Educational Training — Those assigned to this group will be given educational materials about IBS and will discuss the reading material with the therapist. The reading topics include information on gut disorders, anatomy and physiology of the gut, assessment procedures, and how to manage IBS symptoms. Sessions will also consist of weekly reviews of daily records and IBS symptoms. The goal of this intervention is to provide educational training about IBS.
  Arms: 3

SUMMARY:
The purpose of this study is to assess the effect of participation in one of the following interventions: (1) IBS Stress Management; (2) IBS Symptom Management; or (3) IBS Educational Training on improving IBS associated symptoms. It is anticipated that this research will provide information on the usefulness of psychological approaches in treating IBS and will help scientists better understand the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome

Exclusion Criteria:

* GI pathology (organic disease) that affects bowel transit
* Co-morbid pain disorders
* Current or recent history (within 24 months) of drug or alcohol abuse
* Clinical evidence (including physical exam, laboratory tests) of significant medical disease that may interfere with the patient successfully completing the trial
* Planned use of drugs or agents that affect GI motility and/or perception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2002-07; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Changes in Symptoms | 14 days

SECONDARY OUTCOMES:
IBS-specific Quality of Life increase | 14 days
IBS-Specific Beliefs and Coping | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Naliboff, PhD, Principal Investigator — University of California Los Angeles, West Los Angeles VA Healthcare System; Michelle G Craske, PhD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Result] Craske MG, Wolitzky-Taylor KB, Labus J, Wu S, Frese M, Mayer EA, Naliboff BD. A cognitive-behavioral treatment for irritable bowel syndrome using interoceptive exposure to visceral sensations. Behav Res Ther. 2011 Jun;49(6-7):413-21. doi: 10.1016/j.brat.2011.04.001. Epub 2011 Apr 19. PMID 21565328
- See also: Related Info — http://uclacns.org